CLINICAL TRIAL: NCT00612105
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Proof-of-Concept Study to Evaluate the Efficacy of Maximally Tolerated Doses of Retigabine vs. Placebo in Reducing the Pain Associated With Post-Herpetic Neuralgia
Brief Title: Safety/Efficacy Study of Retigabine vs. Placebo in Post-Herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRX-RET-E22-NP201
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic Neuralgia, PHN, Shingles,
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Retigabine
  Interventions: Drug: Retigabine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retigabine — 150mg/day up to 900mg/day
  Arms: 1
Drug: Placebo — daily
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficacy of retigabine vs. placebo in reducing pain associated with post-herpetic neuralgia.

DETAILED DESCRIPTION:
This is a Phase 2a proof of concept study evaluating the safety/efficacy of retigabine vs. placebo in patients with post-herpetic neuralgia. After screening, patients will enter a maximum 6 week titration period followed by a 4 week maintenance period and a 3 week taper phase.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Male or female subjects
* 18-85 years of age
* PHN for more than 6 months after the healing of herpes zoster skin rash
* Has a pain score at screening and randomization that qualifies

Exclusion Criteria:

* Other significant pain that may potentially confound PHN pain assessment
* Previous neurolytic or neurosurgical therapy for PHN
* Subject has evidence of a progressive central nervous system (CNS) disease (e.g. CNS lupus, tumors, multiple sclerosis, Alzheimer's), lesion, or encephalopathy
* Significant psychiatric or neuropsychiatric disorders including but not limited to severe depression, bipolar disorder or schizophrenia spectrum disorder, history of suicide attempt, or recent history of suicidal ideation
* Has clinically significant abnormalities on physical examination, vital signs, ECG, or laboratory tests at the screening visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lineberry, Study Director — Sponsor GmbH
Locations (43):
- United States (39):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Garden Grove, California
  - La Jolla, California
  - San Diego, California
  - Westlake Village, California
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Evansville, Indiana
  - Overland Park, Kansas
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Bay City, Michigan
  - Detroit, Michigan
  - Hattiesburg, Mississippi
  - St Louis, Missouri
  - Toms River, New Jersey
  - New York, New York
  - Raleigh, North Carolina
  - Tabor City, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Mogadore, Ohio
  - Allentown, Pennsylvania
  - Bridgeville, Pennsylvania
  - Charleston, South Carolina
  - Little River, South Carolina
  - North Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Midvale, Utah
- South Africa (4):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Free State
  - Belville, Western Cape
  - George, Western Cape

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Retigabine: Arm Description: Participants started on a total daily dose of 150 milligrams (mg) and were titrated to their maximum tolerated dose (MTD) up to a maximum of 900 mg daily using retigabine 50 mg and/or 100 mg tablets. The dose was increased by 150 mg each week and administered 3 times daily (TID) in equally divided doses. In the Maintenance Phase, retigabine was administered in equally divided doses to maintain the participant's MTD. Participants with moderate to severe side effects during the first week at their MTD and who had attained at least dose level 3 (450 mg) were allowed a one level dose reduction (150 mg). Participants unable to maintain the MTD discontinued the medication. In the Taper Phase, the dose was reduced by one-third during each of the first two weeks, and the study medication was stopped by the third week during the 3-week duration.
- 2: Placebo: Arm Description: Matching placebo tablets of dummy strengths of 50 mg and 100 mg were administered orally TID for up to 6 weeks of the Titration Phase, 4 weeks of the Maintenance Phase, and 3 weeks of the Taper Phase.
Period: Period Title 1: 6-Week Titration Phase
Arm/Group | 1: Retigabine | 2: Placebo
Started | 125 | 62
Completed | 89 | 57
Not Completed | 36 | 5
Not completed — Adverse Event | 18 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Missed study drug for more than two days | 3 | 1
Not completed — Lack of Efficacy | 5 | 0
Not completed — Other | 0 | 1
Period: Period Title 2: 4-Week Maintenance Phase
Arm/Group | 1: Retigabine | 2: Placebo
Started | 89 | 57
Completed | 78 | 55
Not Completed | 11 | 2
Not completed — Adverse Event | 9 | 1
Not completed — Missed study drug for more than two days | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Period Title 3: 3-Week Taper Phase
Arm/Group | 1: Retigabine | 2: Placebo
Started | 86 (Includes participants who discontinued during the titration phase and entered taper phase.) | 58 (Includes participants who discontinued during the titration phase and entered taper phase.)
Completed | 85 | 58
Not Completed | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Retigabine | 2: Placebo | Total
Number analyzed (Participants) | 125 | 62 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 34 | 98
  >=65 years | 61 | 28 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.07) | 61.2 (14.28) | 62.5 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 36 | 100
  Male | 61 | 26 | 87
Region of Enrollment [Number; unit: participants]
  United States | 94 | 47 | 141
  South Africa | 31 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint Will be the Change From Baseline in Average Pain Score Over the Last 7 Days of the Maintenance Phase.
Description: Change from Baseline (BL) was calculated as the value of the average diary pain score for the last 7 days of the MP minus the value of the average pain score at BL (post wash-out period, including the average of the last 7 available entries prior to/including the diary pain measurement on Titration Day 0). Based on their pain experienced during the previous 24 hours, participants assessed their pain every evening at bedtime in an electronic diary by choosing the appropriate number on an 11-point Numerical Rating Scale (NRS): 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain.
Time Frame: Baseline and Week 4 (Maintenance Phase-MP)
Population: Per Protocol (PP) Population: all randomized participants who completed the Titration Phase, had at least 1 dose of treatment in the MP, had at least 3 diary entries in the MP, and did not have any protocol violations or any major protocol deviations
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 81 | 51
Scores on a scale | -2.65 (0.354) | -2.22 (0.387)
Statistical Analysis 1: Comparison: 1: Retigabine vs 2: Placebo; Test type: Superiority or Other; p = 0.2537, ANCOVA; Mean Difference (Net) = -0.43, 95% CI 2-sided [-1.171 to 0.312]

2. Secondary Outcome: Change From Baseline to Weeks 2 and 4 of the Maintenance Phase in Mean In-clinic Pain Assessment
Description: Participants rated their pain during the previous 24 hours at all clinic visits using an 11-point Numerical Rating Scale (NRS): 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain (10=worst possible pain). Change in In-clinic Pain Assessment was calculated by subtracting the average score on the NRS at Week 2 and Week 4 (values for each week were observed cases) of the MP from the average score on the NRS at Baseline (the last non-missing measurement prior to taking study drug).
Time Frame: Baseline and Weeks 2 and 4 (Maintenance Phase - MP)
Population: Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of study medication and had at least one post-randomization efficacy assessment. All participants providing data for the measure are included in the analysis. Differences from the overall population numbers are due to missing data or to subjects missing visits.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 88 | 57
Scores on a scale
  Category Title 1:Week 2; n=88, 57 | -2.7 (2.51) | -2.4 (2.18)
  Category Title 2: Week 4, n=82, 56 | -2.9 (2.41) | -2.4 (2.14)

3. Secondary Outcome: Number of Rescue Medication Tablets Taken Per Day During the Maintenance Phase (MP)
Description: Participants recorded the number of acetaminophen tablets taken during the previous 24 hours in a participant diary. Rescue medication was summarized as the mean number of doses taken per day during each week of the Maintenance Phase (MP) and the mean number of doses taken during all MP weeks.
Time Frame: Weeks 1, 2, 3, and 4 Maintenance Phase
Population: ITT Population. All participants providing data for the measure are included in the analysis. Differences from the overall population numbers are due to missing data or to subjects missing visits.
Measure: Mean (Standard Deviation); unit: Tablets/Day
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 88 | 57
Tablets/Day
  Category Title 1: Week 1; n=88, 57 | 0.92 (1.357) | 0.84 (1.239)
  Category Title 2: Week 2; n=86, 56 | 0.89 (1.228) | 0.79 (1.158)
  Category Title 3: Week 3; n=82, 56 | 0.74 (1.174) | 0.85 (1.254)
  Category Title 4: Week 4; n=76, 55 | 0.83 (1.340) | 0.77 (1.218)
  Category Title 5: All Maintenance Phase Weeks; n=8 | 0.87 (1.211) | 0.83 (1.193)

4. Secondary Outcome: Change From Baseline in Pain Intensity Score at Each Week During the Maintenance Phase (MP)
Description: Least square mean (LSM) of pain intensity was calculated from the NRS score entered by the participants in their diaries at each week during the MP. Participants rated their pain during the previous 24 hours at all clinic visits using an NRS: 0, no pain; 1-3, mild; 4-6, moderate; 7-10 (worst possible pain), severe pain. Change from Baseline was calculated by subtracting the value of the average of the LSM of the NRS score at each week during the MP (the last 7 available diary entries in the MP were used, provided at least 3 existed) from the average Baseline value of the LSM of the NRS score.
Time Frame: Baseline and Weeks 1, 2, 3, and 4 (MP)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 88 | 57
Scores on a scale
  Category Title 1: Week 1; n=88, 57 | -2.35 (0.323) | -2.08 (0.356)
  Category Title 2: Week 2; n=86, 56 | -2.64 (0.337) | -2.34 (0.372)
  Category Title 3: Week 3; n=78, 56 | -2.82 (0.335) | -2.43 (0.363)
  Category Title 4: Week 4; n=75, 55 | -2.82 (0.320) | -2.47 (0.348)

5. Secondary Outcome: Number of Participants Classified as Responders, With a 50% and 30% Pain Reduction From Baseline to the Last 7 Days of the Maintenance Phase
Description: Responders were defined as participants achieving a mean >=50% or >=30% pain reduction based on the NRS score from Baseline to the last 7 days of the MP. Those participants who did not have at least 3 diary entries in the MP, those who withdrew during the Titration Phase (TP), and non-completers (NC: who did not complete the study) were classified as non-responders. The number of responders and responders including non-completers from Baseline to the last 7 days of the MP were reported.
Time Frame: Baseline and Week 4 Maintenance Phase (MP)
Population: ITT Population. All participants providing data for this analysis had to have 7 available baseline diary entries.
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 123 | 61
Participants
  Responders with>=50% Pain Reduction | 33 | 22
  Responders with >=30% Pain Reduction | 52 | 32
  Responders plus NC with>=50% Pain Reduction | 33 | 22
  Responders plus NC with>=30% Pain Reduction | 49 | 31

6. Secondary Outcome: Change From Baseline to the End of the MP (Included All Participants Who Completed Week 4 of the MP and Who Terminated Early During the MP) in Medical Outcomes Study (MOS) Sleep Scale Scores
Description: Change from BL (average value of MOS Sleep Scale score including Overall Sleep Problem [OSP] Index at end of MP minus average BL value) to the end of the MP was summarized for the OSP Index, in addition to the following subscales of the MOS Sleep Scale: Sleep Disturbance; Sleep Adequacy; Snoring; Awakening with Shortness of Breath or with a Headache; Somnolence; and Optimal Sleep. Each item was transformed to a scale with a range of 0-100. For each subscale, except Optimal Sleep, higher scores indicate a greater level of what was being measured (i.e., more snoring, more sleep adequacy, etc.).
Time Frame: Baseline and End of Maintenance Phase (MP) (Week 4).
Population: ITT Population includes all participants who entered MP and provided data. End of Maintenance Phase includes participants who completed Week 4 of the MP and who terminated early during the MP.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Scores on a scale
  Category Title 1: Overall Sleep Problem Index | -5.70 (15.969) | -6.88 (16.814)
  Category Title 2: Sleep Disturbance | -11.47 (21.802) | -9.43 (22.537)
  Category Title 3: Sleep Adequacy | 9.05 (25.536) | 5.26 (26.599)
  Category Title 4: Snoring | 0.7 (23.12) | -2.5 (21.07)
  Title 4:Awaken Short of Breath or with a Headache | -4.8 (19.54) | -4.6 (22.68)
  Category Title 6: Somnolence | 8.10 (20.777) | -3.39 (18.349)

7. Secondary Outcome: Change From Baseline to the End of the MP (Included All Participants Who Completed Week 4 of the MP and Who Terminated Early During the MP) in Sleep Quantity
Description: Change from Baseline in sleep quantity was calculated by subtracting the average value of sleep quantity, calculated in hours, at the end of the MP from the average Baseline value.
Time Frame: Baseline and End of Maintenance Phase (MP) (Week 4).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Hours | 0.5 (1.73) | 0.2 (1.07)

8. Secondary Outcome: Number of Participants With the Indicated Change From Baseline to the End of the Maintenance Phase in Optimal Sleep Based on the Sleep Quantity Domain of the MOS Sleep Scale
Description: Optimal Sleep was based on the Sleep Quantity domain of the MOS Sleep Scale and included the options of "Yes" if sleep quantity was 7-8 hours, and "No" otherwise. "Improved" indicated a change in response of no at baseline to yes at the end of the MP, "Same" indicated no change in response, and "Worse" indicated a change in response from yes at baseline to no at the end of the MP.
Time Frame: Baseline and End of Maintenance Phase (MP) (Week 4).
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Participants
  Category Title 1: Improved | 12 | 8
  Category Title 2: Same | 63 | 42
  Category Title 3: Worse | 9 | 7

9. Secondary Outcome: Number of Participants With the Indicated Overall Patient Global Impression of Change (PGIC)
Description: For the PGIC assessment, participants were asked to assess their overall status since they initiated the study drug to the end of the Maintenance Phase using a 7-point categorical scale: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. All participants who completed Week 4 of the Maintenance Phase and participants who terminated early during the Maintenance Phase were assessed.
Time Frame: Baseline to the end of Maintenance Phase (MP) (Week 4)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Participants
  Category Title 1: Very Much Improved | 20 | 8
  Category Title 2: Much Improved | 27 | 15
  Category Title 3: Minimally Improved | 19 | 10
  Category Title 4: No Change | 14 | 21
  Category Title 5: Minimally Worse | 3 | 2
  Category Title 6: Much Worse | 1 | 1
  Category Title 7: Very Much Worse | 0 | 0

10. Secondary Outcome: Mean Score on the Treatment Satisfaction Questionnaire for Medication (TSQM) at the End of the Maintenance Phase
Description: The TSQM assessed the participant's overall satisfaction with treatment, including subscales to assess effectiveness, side effects, convenience, and global satisfaction. Raw scores from the scale were transformed into a numeric scale ranging from 0 to 100, where higher scores indicated greater satisfaction with treatment. TSQM was reported at the end of the MP. Participants who completed Week 4 of the MP and who terminated early during the MP were assessed.
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: ITT Population includes all participants who entered MP and provided data. End of Maintenance Phase includes participants who completed Week 4 of the MP and who terminated early during the MP. Differences from the overall population numbers are due to missing data or to participants missing visits.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Scores on a scale
  Category Title 1: Effectiveness; n=83, 57 | 59.10 (29.392) | 49.51 (30.143)
  Category Title 2: Side Effects; n=82, 57 | 67.76 (28.097) | 92.11 (18.280)
  Category Title 3: Convenience; n=84, 57 | 69.97 (21.423) | 74.66 (19.782)
  Category Title 4: Global Satisfaction; n=84, 57 | 58.67 (30.649) | 52.88 (34.517)

11. Secondary Outcome: Scores on the Brief Pain Inventory-Short Form (BPI-SF) at the End of the MP for All Participants Who Completed Week-4 of the MP and Who Terminated Early During the MP
Description: The BPI-SF assessed pain intensity, pain relief from medication, and pain interference with function over the previous 24 hours. Pain intensity was assessed by the mean of 4 intensity items rated on a 0-10 categorical scale: 0=no pain, 10=pain as bad as you can imagine. Pain interference was assessed by determining the mean of the 7 interference items on a 0-10 categorical scale ranging from 0=does not interfere to 10=completely interferes. The level of pain relief provided by treatment was assessed on an 11-point categorical scale ranging from 0% to 100%
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Scores on a scale
  Category Title 1: Pain Intensity; n=74, 49 | 3.17 (2.092) | 3.58 (2.299)
  Category Title 2: Pain Interference; n=75, 49 | 2.00 (2.159) | 2.27 (2.147)
  Category Title 3: Pain Relief; n=74, 48 | 58.4 (35.04) | 49.4 (36.17)

12. Secondary Outcome: Scores on the Medical Outcomes Short Form-36 (SF-36) at the End of the MP for All Participants Who Completed Week 4 of the MP and Who Terminated Early During the MP
Description: Least square (LS) mean calculated based on participant's assessment of SF-36,a quality of life questionnaire consisting of 36 items grouped into 8 domains. These 8 domains further grouped into 2 overall summary measures,physical health and mental health. Higher scores on SF-36 represented better state of health. Physical/mental components summarized the data of all the physical/mental domains of SF-36 and higher scores represented better state of health.
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 55
Scores on a scale
  Category Title 1: General health; n=83, 55 | 51.12 (0.816) | 50.47 (1.002)
  Category Title 2: Physical Functioning; n=84, 55 | 43.82 (0.870) | 45.54 (1.076)
  Category Title3: Role limitations, physical; n=84, | 43.22 (1.046) | 43.30 (1.293)
  Category Title4: Role limitations, emotional; n=84 | 44.31 (1.226) | 42.68 (1.517)
  tegory Title 5: Social Functioning; n=84, 55 | 50.14 (0.858) | 50.25 (1.061)
  Category Title 6: Bodily Pain; n=84, 55 | 47.23 (0.883) | 45.60 (1.091)
  Category Title 7: Vitality; n=84, 55 | 51.68 (0.904) | 53.94 (1.117)
  Category Title 8: Mental Health; n=84, 55 | 51.66 (0.871) | 51.34 (1.076)
  Category Title9: Physical Component Summary; n=83, | 45.26 (0.691) | 45.65 (0.849)
  Category Title10: Mental Component Summary; n=83, | 51.22 (0.944) | 50.91 (1.160)

13. Secondary Outcome: Scores for Reported Health Transition at the End of the MP for All Participants Who Completed Week 4 of the MP and Who Terminated Early During the MP
Description: The least square (LS) mean score for reported health transition was calculated based on the scores (ranging from 1 to 5) given by the participant in answer to the following question: "Compared to 1 year ago, how would you rate your health in general now?". Lower numbers represent a better state of health.
Time Frame: End of maintenance Phase (MP) (Week 4)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 83 | 55
Scores on a scale | 2.68 (0.102) | 2.37 (0.125)

14. Secondary Outcome: Number of Participants With the Indicated Responses at Baseline to the Question: "How Painful Was the Affected Side Compared to the Opposite Side?" in an Assessment of Tactile Allodynia
Description: At Baseline, the investigator conducted the Neuropathic Pain Physical Examination (NPPE) to examine hyperalgesia and allodynia (tactile and cold). Tactile allodynia was assessed with a foam brush, based on the question:"How painful was the affected side compared to the opposite side?".
Time Frame: Baseline Phase (Day -7 to Randomization Day 0)
Population: ITT Population - All participants providing data for the measure are included in the analysis. Differences from the overall population numbers are due to missing data or to subjects missing visits.
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 124 | 61
Participants
  Category Title 1: More Painful | 89 | 40
  Category Title 2: The Same | 19 | 14
  Category Title 3: Less Painful | 16 | 7

15. Secondary Outcome: Number of Participants With the Indicated Responses at Baseline to the Questions of "Is it Cool?" and "Is it Painful?" in an Assessment of Cold Threshold and Allodynia
Description: At Baseline the investigator conducted the NPPE to examine hyperalgesia and allodynia (tactile and cold). Cold threshold and allodynia was assessed to determine if a metal bar felt cool and if it felt painful, based on the questions:"Is it cool?" and "Is it painful?"
Time Frame: Timeframe: Baseline Phase (Day -7 to Randomization Day 0)
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 124 | 61
Participants
  Is Not Cool | 19 | 9
  Is Cool | 105 | 52
  Is Not Painful | 67 | 34
  Is Painful | 57 | 27

16. Secondary Outcome: Number of Subjects With the Indicated Responses at Baseline to the Questions: "How Sharp Was the Affected Side Compared to the Opposite Side?" and "How Painfule Was the Affected Side Compared to the Opposite Side?" in an Assessment of Hyperalgesia
Description: At Baseline the investigator conducted the NPPE to examine hyperalgesia and allodynia (tactile and cold). Hyperalgesia is defined as increased sensitivity to pain, which may be caused by damage to peripheral nerves. It was assessed with a pinprick brush, based on the questions: "How sharp was the affected side compared to the opposite side?" and "How painfule was the affected side compared to the opposite side?"
Time Frame: Baseline Phase (Day -7 to Randomization Day 0)
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 124 | 61
Participants
  More Sharp | 66 | 32
  The Same(sharp) | 7 | 10
  Less sharp | 51 | 19
  More Painful | 71 | 38
  The Same(pain) | 19 | 7
  Less Painful | 34 | 16

17. Secondary Outcome: Number of Participants With the Indicated Responses at the End of the MP to the Question: "How Painful Was the Affected Side Compared to the Opposite Side?" in an Assessment of Tactile Allodynia
Description: At the end of the MP, the investigator conducted the NPPE (an examination of the effect of retigabine on sensory abnormalities) to examine hyperalgesia and allodynia (tactile and cold). Tactile allodynia was assessed with a foam brush, based on the question:"How painful was the affected side compared to the opposite side?" End of Maintenance Phase includes participants who completed Week 4 of the MP and who terminated early during the MP.
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Participants
  More Painful | 30 | 29
  The Same | 44 | 20
  Less Painful | 10 | 8

18. Secondary Outcome: Number of Participants With the Indicated Responses at the End of the MP to the Questions of "Is it Cool?" and "Is it Painful?" in an Assessment of Cold Threshold and Allodynia
Description: At the end of the MP, the investigator conducted the NPPE (an examination of the effect of retigabine on sensory abnormalities) to examine hyperalgesia and allodynia (tactile and cold). Cold threshold and allodynia was assessed to determine if a metal bar felt cool and if it felt painful, based on the questions:"Is it cool?" and "Is it painful?"
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Participants
  Is Not Cool | 14 | 7
  Is Cool | 70 | 50
  Is Not Painful | 63 | 44
  Is Painful | 21 | 13

19. Secondary Outcome: Number of Participants With Indicated Responses at the End of the MP to the Questions: "How Sharp Was the Affected Side Compared to the Opposite Side?" and "How Painful Was the Affected Side Compared to the Opposite Side?" in an Assessment of Hyperalgesia
Description: At the end of the MP, the investigator conducted the NPPE (an examination of the effect of retigabine on sensory abnormalities) to examine hyperalgesia and allodynia (tactile and cold). Hyperalgesia is defined as increased sensitivity to pain, which may be caused by damage to peripheral nerves. It was assessed with a pinprick brush, based on the questions:"How sharp was the affected side compared to the opposite side?" and How painful was the affected side compared to the opposite side?"
Time Frame: End of Maintenance Phase (MP) (Week 4)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 84 | 57
Participants
  More Sharp | 29 | 24
  The Same(sharp) | 24 | 19
  Less Sharp | 31 | 14
  More Painful | 31 | 24
  The Same(pain) | 28 | 18
  Less Painful | 25 | 15

20. Secondary Outcome: Change From Baseline in the Average Diary Pain Score to the Last 7 Days of the Maintenance Phase by Post Herpetic Neuralgia (PHN) Subtype "Irritable Nociceptors"
Description: Participants were stratified into four different PHN subtypes based on the NPPE. Participants with pain, abnormal sensitization of the specific receptor (irritable nociceptors), and with minimal sensory loss were stratified in the"irritable nociceptors" subtype. Based on their pain experienced during the previous 24 hours, participants assessed their pain every evening at bedtime in an electronic diary by choosing the appropriate number on an 11-point NRS: 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain.
Time Frame: Baseline and Week 4 Maintenance Phase (MP)
Population: ITT Population. Only participants in the specified subgroup were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 17 | 13
Scores on a scale | -1.78 (2.166) | -2.85 (2.163)

21. Secondary Outcome: Change From Baseline in the Average Diary Pain Score to the Last 7 Days of the Maintenance Phase by Post Herpetic Neuralgia (PHN) Subtype"Deafferentation Type 1 (D Type 1)"
Description: Participants stratified into 4 different PHN subtypes based on NPPE. Participants with marked sensory loss associated with severe burning pain upon slight mechanical stimuli (allodynia) were stratified in the "deafferentation type 1" subtype. Based on their pain experienced during the previous 24 hours, participants assessed their pain every evening at bedtime in an electronic diary by choosing the appropriate number on an 11-point NRS: 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain.
Time Frame: Baseline and Week 4 Maintenance Phase (MP)
Population: ITT Population. Only participants in the specified subgroup were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 4 | 2
Scores on a scale | -3.57 (2.368) | -5.29 (0.000)

22. Secondary Outcome: Change From Baseline in the Average Diary Pain Score to the Last 7 Days of the Maintenance Phase by Post Herpetic Neuralgia (PHN) Subtype "Deafferentation Type 2 (D Type 2)"
Description: Participants stratified into 4 different PHN subtypes based on NPPE. Participants with marked sensory loss and severe spontaneous burning pain without allodynia associated with reorganization of central nerve fibers were stratified in the "deafferentation type 2" subtype. Based on their pain experienced during the previous 24 hours, participants assessed their pain every evening at bedtime in an electronic diary by choosing the appropriate number on an 11-point NRS: 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain.
Time Frame: Baseline and Week 4 Maintenance phase (MP)
Population: ITT Population. Only participants in the specified subgroup were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 4 | 2
Scores on a scale | -4.14 (0.00) | 0.00 (0.00)

23. Secondary Outcome: Change From Baseline in the Average Diary Pain Score to the Last 7 Days of the Maintenance Phase by Post Herpetic Neuralgia (PHN) Subtype "Unclassifiable"
Description: Participants stratified into 4 different PHN subtypes based on NPPE. Participants who could not be specifically differentiated in any of the other three subtypes were stratified as "unclassifiable" meaning that the participants could not be classified into any of the predefined PHN subtypes. Based on their pain experienced during the previous 24 hours, participants assessed their pain every evening at bedtime in an electronic diary by choosing the appropriate number on an 11-point NRS: 0, no pain; 1 to 3, mild; 4 to 6, moderate; 7 to 10, severe pain.
Time Frame: Baseline and Week 4 Maintenance Phase (MP)
Population: ITT Population. Only participants in the specified subgroup were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1: Retigabine | 2: Placebo
Number analyzed (Participants) | 66 | 42
Scores on a scale | -2.69 (2.285) | -1.87 (1.870)

ADVERSE EVENTS:
Description: SAEs and AEs are reported for all Phases (Titration, Maintenance and Taper).
Arm/Group | 1: Retigabine | 2: Placebo
Serious Adverse Events (participants affected / at risk) | 7/125 | 1/62
Other Adverse Events (participants affected / at risk) | 98/125 | 29/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1: Retigabine (N=125) | 2: Placebo (N=62)
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Maculopathy (Eye disorders) | 1 | 0
Retinal Detatchment (Eye disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulmonaryy Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1: Retigabine (N=125) | 2: Placebo (N=62)
Dizziness (Nervous system disorders) | 45 | 8
Somnolence (Nervous system disorders) | 41 | 7
Headache (Nervous system disorders) | 23 | 8
Memory Impairment (Nervous system disorders) | 9 | 0
Amnesia (Nervous system disorders) | 7 | 0
Paraesthesia (Nervous system disorders) | 7 | 0
Nausea (Gastrointestinal disorders) | 15 | 3
Diarrhea (Gastrointestinal disorders) | 12 | 6
Dry Mouth (Gastrointestinal disorders) | 9 | 2
Confusional State (Psychiatric disorders) | 9 | 1
Fatigue (General disorders) | 13 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Urinary Tract Infection (Infections and infestations) | 8 | 4
Vision Blurred (Eye disorders) | 8 | 3
Vertigo (Ear and labyrinth disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Valeant supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial